CLINICAL TRIAL: NCT01779336
Title: An Open Label Multicentre Phase 1 Study of Oral IGF-1R Inhibitor PL225B in Subjects With Advanced Refractory Solid Tumors.
Brief Title: Clinical Study of Oral IGF-1R Inhibitor in Subjects With Advanced Refractory Solid Tumors
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision not related to patient safety
Sponsor: Piramal Enterprises Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PL225B/71/11
Record Dates: First submitted 2013-01-28; First posted 2013-01-30 (Estimated); Last update posted 2014-09-29 (Estimated); Status verified 2014-09

CONDITIONS: Advanced Refractory Solid Tumors
Keywords: Advanced Refractory Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PL225B (Experimental): Patients will receive study drug on a daily basis until disease progression or unacceptable toxicity in sequential cohorts following accelerated titration design.
  Interventions: Drug: PL225B

INTERVENTIONS:
Drug: PL225B — * Patients will receive study drug on a daily basis for twenty-one (21) days according to the dose and schedule specified for a particular cohort of therapy.
  * This 21 day administration will define a treatment cycle.
  * Patients may receive consecutive treatment cycles until evidence of disease progression, intolerance of therapy, or withdrawal from the protocol as specified.

SUMMARY:
Clinical study of oral IGF-1R inhibitor PL225B in subjects with advanced refractory solid tumors. The primary objective is to determine the maximum tolerated dose and dose limiting toxicity (ies) of oral IGF-1R inhibitor PL225B in subjects with advanced refractory solid tumors.

DETAILED DESCRIPTION:
An open label multicentre Phase 1 study of oral IGF-1R inhibitor PL225B in subjects with advanced refractory solid tumors. This is a dose-finding trial using the modified Accelerated Titration Design with 3 new subjects per cohort and 100% dose increments in the accelerated phase followed by standard phase with 40% dose increments.Subjects will receive study drug on a daily basis for twenty-one (21) days according to the dose and schedule specified for a particular cohort of therapy. Toxicity profile of the drug will be assessed during Cycle 1 of subject treatment in each cohort for determination of Maximum Tolerated Dose (MTD) according to the schedule given below.

ELIGIBILITY:
Inclusion Criteria:

* Subjects having histologically and/or cytologically confirmed non-haematological malignancy that is metastatic or unresectable and for which standard curative or palliative treatment does not exist or is no longer effective
* Subjects should have measurable or evaluable disease
* Subjects of either sex, of all races and ethnic groups, and ≥18 years of age
* ECOG (Eastern Cooperative Oncology Group) performance status 0-1
* Subjects with life expectancy of at least 4 months
* Subjects with fasting plasma glucose ≤ 125 mg/dL and HbA1c < 6.5 % at screening Subjects with fasting plasma glucose ≤150 mg/dL and HbA1c ≤ 7.0 % at screening for the Diabetes Expansion Cohort.
* For the Diabetes Expansion Cohort - Subjects with known history of type 2 diabetes mellitus that are well-controlled on a stable dose of oral anti-diabetic agents such as metformin and/or sulfonylureas for 4 weeks prior to screening.
* Subjects must have normal organ and marrow function as defined below:

  1. Absolute neutrophil count ≥ 1500/cmm
  2. Platelets ≥ 100,000/cmm
  3. Total bilirubinwithin normal limits of the institution
  4. AST/ALT ≤ 2.5 X institutional upper limit of normal (ULN) or ≤ 5 X institutional upper limit of normal (ULN) in the presence of liver metastases
  5. Creatinine ≤ 1.5 X institutional upper limit of normal (ULN)
* Subjects willing for repeat oral dosing and follow-up, including pharmacokinetic sampling
* Women of childbearing potential and men willing to agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, during the duration of study participation and for at least 4 weeks after withdrawal from the study, unless they are surgically sterilised
* Ability to understand and the willingness to provide a written informed consent document

Exclusion Criteria

* Subjects who have received any prior chemotherapy, radiotherapy, biologic/targeted anti-cancer therapy or surgery within 4 weeks (6 weeks for monoclonal antibodies, radioactive monoclonal antibodies or any radio- or toxin- immunoconjugates) before the first study drug administration and have not recovered (to AEs < Grade 2) from the toxic effects from any prior therapy
* Subjects having received any other investigational agents within 4 weeks prior to the first study drug administration and have not recovered completely (to AEs < Grade 2) from the side effects of the earlier investigational agent
* Subjects with documented history of diabetes mellitus except for the Diabetes Expansion Cohort
* For the Diabetes Expansion Cohort - Subjects who have type 1 diabetes mellitus, maturity onset diabetes of the young, hyperglycemia due to reasons other than type 2 diabetes mellitus.
* For the Diabetes Expansion Cohort - Subjects who currently require insulin, thiazolidinediones, dual proliferator-activated receptors (PPAR) agonists, glucagon-like peptide (GLP-1) analogues, dipeptidyl peptidase (DPP-IV) inhibitors or have received the same in the 4 weeks prior to screening.
* Subjects with known complications of diabetes like diabetic nephropathy or diabetic retinopathy
* Subjects with known brain metastases
* Subjects with gastrointestinal abnormalities including inability to take oral medication, malabsorption or other conditions like chronic inflammatory bowel disease that may affect absorption.
* Subjects with a history of myocardial infarction or uncontrolled cardiac dysfunction during the previous 6 months
* Subjects with baseline QTc interval >470 msec at screening
* Subjects on warfarin. Prophylactic anticoagulation with low molecular weight heparin is allowed
* Subjects with history of anaphylaxis or angioedema, bronchial asthma, peptic ulcer and clinically significant food or drug allergy
* Subjects with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Women who are pregnant or nursing
* Subjects with known seropositivity to human immunodeficiency virus (HIV), positive for Hepatitis B, positive for Hepatitis C (antigen positive), or known hepatic cirrhosis

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2012-12; Primary Completion 2014-11 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose | End of Cycle 1 (i.e. 21 Days)
  Subjects will receive study drug on a daily basis for twenty-one (21) days according to the dose and schedule specified for a particular cohort of therapy.Toxicity profile of the drug will be assessed during Cycle 1 of subject treatment in each cohort for determination of Maximum Tolerated Dose (MTD).

SECONDARY OUTCOMES:
Number of subject with adverse events | Until disease progression or unacceptable toxicity (expected to be 4-6 months)
  The toxic effects of the drug would be assessed from adverse events, vital signs and by clinically significant changes in the laboratory evaluations.
Pharmacokinetic profile(Cmax,Tmax and AUC) | Until disease progression or unacceptable toxicity (expected to be 4-6 months)
  The following PK parameters will be calculated: Cmax (peak plasma concentration), Tmax (time to peak plasma concentration), AUC0-t (area under the plasma concentration curve from time zero to time of last quantifiable concentration), AUC0-12, AUC0-inf (area under the plasma concentration curve from time zero extrapolated to infinity), percent AUC extrapolated, kel (elimination rate constant), t1/2 (elimination half-life), CL/F (oral clearance), Vz/F (oral apparent volume of distribution) and Racc (accumulation ratio).
Activity of PL225B based on selected biomarkers | Until disease progression or unacceptable toxicity (expected to be 4-6 months)
  Plasma samples will be used for analysis of circulating exploratory biomarkers which are likely to change in response to PL225B administration.
Objective response | Until disease progression or unacceptable toxicity (expected to be 4-6 months)
  Evaluation of Response: Clinical responses will be presented patient wise for different dose levels.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Anthony El-Khoueiry, MD, Principal Investigator — University of Southern California
Locations (5):
- USC Norris Comprehensive Cancer Center, Los Angeles, California, United States
- India (4):
  - Central India Cancer Research Institute, Nagpur, Maharashtra
  - Curie Manavata Cancer Centre, Nashik, Maharashtra
  - Ruby Hall Clinic, Pune, Maharashtra
  - Meenakshi Mission Hospital and Research Centre, Madurai, Tamil Nadu